CLINICAL TRIAL: NCT05997836
Title: Behavioral Health Interdisciplinary Program - Collaborative Chronic Care Model (BHIP-CCM) Enhancement Project 2.0 (QUE 20-026)
Brief Title: Behavioral Health Interdisciplinary Program - Collaborative Chronic Care Model (BHIP-CCM) Enhancement Project 2.0
Acronym: BHIP-CCM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs Office of Mental Health and Suicide Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 23-002
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Mental Health
Keywords: collaborative care
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study will use a stepped wedge design, with participating medical centers assigned to one of four different waves. Wave 1 will begin the trial receiving implementation facilitation. Waves 2-4 will begin the trial receiving centralized technical assistance, and will then cross over to implementation facilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Wave 1 (Other): Study design is a stepped wedge; Wave 1 begins by receiving Implementation Facilitation
  Interventions: Other: Implementation Facilitation
- Wave 2 (Other): Study design is a stepped wedge; Wave 2 begins by receiving Centralized Technical Assistance before crossing over to Implementation Facilitation
  Interventions: Other: Implementation Facilitation; Other: Centralized Technical Assistance
- Wave 3 (Other): Study design is a stepped wedge; Wave 3 begins by receiving Centralized Technical Assistance before crossing over to Implementation Facilitation
  Interventions: Other: Implementation Facilitation; Other: Centralized Technical Assistance
- Wave 4 (Other): Study design is a stepped wedge; Wave 4 begins by receiving Centralized Technical Assistance before crossing over to Implementation Facilitation
  Interventions: Other: Implementation Facilitation; Other: Centralized Technical Assistance

INTERVENTIONS:
Other: Implementation Facilitation — Implementation Facilitation involves and External Facilitator (from outside of the participating medical center) and an Internal Facilitator (from inside the participating medical center) working together to help BHIP teams within the site adopt care practices that are more consistent with the CCM
  Other Names: IF
Other: Centralized Technical Assistance — Centralized Technical Assistance involves having external experts available for ad hoc consultation related to collaborative BHIP care practices.
  Other Names: CTA
  Arms: Wave 2; Wave 3; Wave 4

SUMMARY:
This quality improvement project aims to help outpatient mental health teams, known as Behavioral Health Interdisciplinary Program (BHIP) teams, adopt more collaborative care practices (consistent with the collaborative chronic care model or CCM). The investigators therefore aim to use two different implementation strategies -- centralized technical assistance and implementation facilitation -- to align BHIP teams' care practices more closely with the principles of the CCM.

DETAILED DESCRIPTION:
This quality improvement project aims to help outpatient mental health teams, known as Behavioral Health Interdisciplinary Program (BHIP) teams, adopt more collaborative care practices (consistent with the collaborative chronic care model or CCM). The investigators therefore aim to use two different implementation strategies -- centralized technical assistance and implementation facilitation -- to align BHIP teams' care practices more closely with the principles of the CCM.

The two primary outcomes of this project are:

1. BHIP team collaboration, as evidenced by improved scores in the Role Clarity and Team Primacy dimensions of the Team Development Measure (TDM)
2. BHIP team clinical effectiveness, as evidenced by reduction in mental health hospitalizations among Veterans treated by the BHIP teams that have received the two types of implementation strategies described above.

ELIGIBILITY:
Inclusion Criteria:

* Note that treatment assignment will be at the facility level, and given the stepped wedge design, sites in Waves 2-4 will cross over from Centralized Technical Assistance to Implementation Facilitation.
* At the provider level (for completing the TDM), the primary inclusion criterion is clinicians working on BHIP Teams at the participating medical centers.
* At the patient level (for mental health hospitalizations, costs, and all-cause mortality), the primary inclusion criterion is Veterans treated by the BHIP teams at the participating medical centers.
* Note that, for mental health hospitalizations, separate sites have been identified as comparators using a balancing algorithm.

Exclusion Criteria:

* Patients with a diagnosis of dementia in the electronic medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81424 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Role Clarity and Team Primacy subdomains of the Team Development Measure (TDM) | Primary comparison will be between pre-implementation facilitation and post-implementation facilitation (8 months after the pre-implementation administration).
  The TDM is a measure of team functioning, and the two listed subdomains represent the co-primary outcome for the study. Note that, due to the stepped wedge design, only Wave 3 and Wave 4 sites will also have a pre-centralized technical assistance administration of the TDM. Also note that the primary time frame for this outcome, as listed above, will be post-implementation facilitation (8 months after the pre-implementation administration). Secondary analysis will also investigate one year post-implementation facilitation (20 months after the pre-implementation administration).
Mental health hospitalization rate among Veterans treated within each BHIP team. | Primary comparison will be between pre-implementation facilitation and post-implementation facilitation (8 months after the pre-implementation administration).
  Mental health hospitalizations represent a measure of clinical effectiveness (co-primary outcome for the study). Note that, due to the stepped wedge design, only Wave 3 and Wave 4 sites will also have a pre-centralized technical assistance calculation of the mental health hospitalization rate. Also note that the primary time frame for this outcome, as listed above, will be post-implementation facilitation (8 months after the pre-implementation administration). Secondary analysis will also investigate one year post-implementation facilitation (20 months after the pre-implementation administration).

SECONDARY OUTCOMES:
Treatment cost | Primary comparison will be between pre-implementation facilitation and post-implementation facilitation (8 months after the pre-implementation administration).
  The investigators will calculate estimated treatment costs for Veterans treated by participating BHIP teams. Note that the primary time frame for this outcome, as listed above, will be post-implementation facilitation (8 months after the pre-implementation administration). Secondary analysis will also investigate one year post-implementation facilitation (20 months after the pre-implementation administration).
All-cause mortality | Primary comparison will be between pre-implementation facilitation and post-implementation facilitation (8 months after the pre-implementation administration).
  The investigators will calculate all-cause mortality for Veterans treated by participating BHIP teams. Note that the primary time frame for this outcome, as listed above, will be post-implementation facilitation (8 months after the pre-implementation administration). Secondary analysis will also investigate one year post-implementation facilitation (20 months after the pre-implementation administration).
Treatment costs and hospitalization data compared to non-intervention sites | Post-facilitation (8 months after start of implementation facilitation) and post-sustainment (12 months after post-facilitation)
  For mental health hospitalization and treatment costs, the investigators will compare results from intervention sites to other sites that did not undergo implementation facilitation (i.e. sites from outside the trial that are similar to intervention sites on variables like facility complexity and urban/rural location).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. Miller, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA; Sara J. Landes, PhD MA BA, Principal Investigator — Central Arkansas Veterans Healthcare System , Little Rock, AR
Locations (17):
- United States (17):
  - Northern Arizona VA Health Care System, Prescott, AZ, Prescott, Arizona
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Fayetteville VA Medical Center, Fayetteville, NC, Fayetteville, North Carolina
  - Jackson C. Montgomery VA Medical Center, Muskogee, OK, Muskogee, Oklahoma
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - West Texas VA Health Care System, Big Spring, TX, Big Spring, Texas
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - Clarksburg Louis A. Johnson VA Medical Center, Clarksburg, WV, Clarksburg, West Virginia
  - Huntington VA Medical Center, Huntington, WV, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No